CLINICAL TRIAL: NCT01762917
Title: Influence of Bag Volume Variation in Inert Gas Rebreathing Pulmonary Blood Flow Measurements on the Reproducibility in Patients With Pulmonary Diseases
Brief Title: Influence of Bag Volume Variation on the Reproducibility of Inert Gas Rebreathing
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Joachim Saur, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: IGR_Vbag_MA
Record Dates: First submitted 2012-12-21; First posted 2013-01-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Bronchial Asthma; Restrictive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Obstruction: Patients suffering from pulmonary obstruction
- Restriction: Patients suffering from pulmonary restriction
- Controls: Pulmonary healthy controls

SUMMARY:
Non-invasive inert gas rebreathing (IGR) based on the Fick Principle showed promising results in the determination of pulmonary blood flow (PBF). The volume of the rebreathing bag (Vbag) is proposed by the system, however, elderly patients or those suffering from high grade pulmonary diseases might be unable to entirely rebreathe this volume and therefore fail to completely mix the test gases. The aim of our study is to evaluate the effect of adapting Vbag on the reproducibility of IGR measurements in patients with obstruction (group A), restriction (group B) and pulmonary healthy controls (group C).

ELIGIBILITY:
Inclusion Criteria:

* ability to perform rebreathing maneuver

Exclusion Criteria:

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: inpatients and outpatients, internal medicine, university hospital
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
pulmonary blood flow | 1 day
  variation of serial pulmonary blood flow measurements

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Mannheim, Mannheim, Germany